CLINICAL TRIAL: NCT05826002
Title: Optimization of a Digital Self-guided Psychological Intervention for Insomnia: A Randomized Factorial Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Martin Kraepelien, Clinical Psychologist, Principal Investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-07226-01
Record Dates: First submitted 2023-03-27; First posted 2023-04-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Insomnia
Keywords: Insomnia; ICBT; Factorial Experiment; Optimization; User Interface; Adaptive Treatment Strategy; Prompts; Digital Intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A 2x2x2 randomized factorial experiment, where adult participants with insomnia get to use a digital self-guided intervention for insomnia. Three factors/treatment features will be manipulated in the experiment, namely: 1) an optimized graphical user interface (yes or no), 2) an adaptive treatment strategy (yes or no), and 3) daily prompts to use the intervention (yes or no). The factorial experiment will create 8 equally large groups (1:1:1:1:1:1:1:1), who will receive the different combinations of features.
Who Masked: Participant
Masking Description: Participants will be blinded to what condition they are randomized to, and will not receive information concerning what features are being manipulated in the experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Digital insomnia intervention (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (no), adaptive treatment strategy (no), daily prompts (no).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + optimized user interface (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (yes), adaptive treatment strategy (no), daily prompts (no).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + adaptive treatment strategy (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (no), adaptive treatment strategy (yes), daily prompts (no).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + optimized user interface, adaptive treatment strategy (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (yes), adaptive treatment strategy (yes), daily prompts (no).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + daily prompts (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (no), adaptive treatment strategy (no), daily prompts (yes).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + optimized user interface, daily prompts (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (yes), adaptive treatment strategy (no), daily prompts (yes).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + adaptive treatment strategy, daily prompts (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (no), adaptive treatment strategy (yes), daily prompts (yes).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia
- Digital insomnia intervention + optimized user interface, adaptive treatment strategy, daily prompts (Active Comparator): This group receives the following combination of treatment features: optimized graphical user interface (yes), adaptive treatment strategy (yes), daily prompts (yes).
  Interventions: Behavioral: Digital self-guided psychological intervention for insomnia

INTERVENTIONS:
Behavioral: Digital self-guided psychological intervention for insomnia — A four week digital self-guided intervention for insomnia, with content derived from Cognitive Behavioral Therapy for insomnia, and with a clinical interview before and after the intervention.

SUMMARY:
In a previous pilot study, a digital self-guided intervention for insomnia showed preliminary positive effects on insomnia symptoms. In order to optimize the digital self-guided format, this study will evaluate the added value of three treatment features on treatment engagement and insomnia symptoms. The participants will be adults with insomnia. The trial will be a 2x2x2 randomized factorial experiment, where the following features/factors will be manipulated: an optimized graphical user interface (yes or no), an adaptive treatment strategy (yes or no), and daily prompts to use the intervention (yes or no). The factorial experiment will create 8 equally large groups (1:1:1:1:1:1:1:1), who will receive the different combinations of features. The main outcome will be the effect on treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. ≥ 15 points on Insomnia Severity Index.
3. Insomnia diagnosis, according to criteria in the Diagnostic and Statistical Manual of mental disorders-5 (somatic/psychiatric comorbidity is allowed).
4. Good understanding of the Swedish language.
5. No practical obstacles to participate in treatment and assessments.
6. Daily access to computer/smart-phone/tablet with Internet access.
7. Can receive phone calls and text messages during the study period.

Exclusion Criteria:

1. Sleep diseases, such as narcolepsy or sleep apnea.
2. Somatic or psychiatric illnesses that either are directly contraindicated for the treatment, require other treatment, or entail symptoms/a functional level making it too difficult to participate in the study.
3. Alcohol/drug abuse, or medication with side effects on sleep (however, sleep medication is allowed).
4. Working nights or night shifts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Engagement with intervention method | Up to 12 months after treatment
  Treatment engagement questionnaire (self-rated study-specific questionnaire), score range 0-21 (0-7 per item), higher is better
Engagement with intervention method | Immediately after treatment (4 weeks after treatment start)
  Treatment engagement questionnaire (self-rated study-specific questionnaire), score range 0-21 (0-7 per item), higher is better

SECONDARY OUTCOMES:
Change in Insomnia symptoms | Change from baseline (right before treatment start) up to 12 months after treatment
  Insomnia Severity Index (self-rated), score range 0-28, lower is better
Change in Insomnia symptoms | Change from baseline (right before treatment start) to immediately after treatment (4 weeks after treatment start)
  Insomnia Severity Index (self-rated), score range 0-28, lower is better
Change in Depression symptoms | Change from baseline (right before treatment start) up to 12 months after treatment
  Patient Health Questionnaire-9 (self-rated), score range 0-27, lower is better
Change in Depression symptoms | Change from baseline (right before treatment start) to immediately after treatment (4 weeks after treatment start)
  Patient Health Questionnaire-9 (self-rated), score range 0-27, lower is better
Change in Anxiety symptoms | Change from baseline (right before treatment start) up to 12 months after treatment
  Generalized Anxiety Disorder-7 (self-rated), score range 0-21, lower is better
Change in Anxiety symptoms | Change from baseline (right before treatment start) to immediately after treatment (4 weeks after treatment start)
  Generalized Anxiety Disorder-7 (self-rated), score range 0-21, lower is better
Change in Life quality | Change from baseline (right before treatment start) up to 12 months after treatment
  Brunnsviken Brief Quality of life scale (self-rated), score range 0-96, higher is better
Change in Life quality | Change from baseline (right before treatment start) to immediately after treatment (4 weeks after treatment start)
  Brunnsviken Brief Quality of life scale (self-rated), score range 0-96, higher is better
Change in Daily function | Change from baseline (right before treatment start) up to 12 months after treatment
  World Health Organization Disability Assessment Schedule (self-rated), score rang 0-100, lower is better
Change in Daily function | Change from baseline (right before treatment start) to immediately after treatment (4 weeks after treatment start)
  World Health Organization Disability Assessment Schedule (self-rated), score rang 0-100, lower is better
Treatment credibility | 2 weeks after treatment start (mid-treatment)
  Credibility/Expectancy Questionnaire (self-rated), score range 0-50, higher is better
Intervention/system usability | 2 weeks after treatment start (mid-treatment)
  System Usability Scale (self-rated), score range 0-100, higher is better
Treatment satisfaction | Immediately after treatment (4 weeks after treatment start)
  Client Satisfaction Questionnaire-8 (self-rated), score range 8-32, higher is better

OTHER OUTCOMES:
Clinician time | Immediately after treatment (4 weeks after treatment start)
  Time in minutes the clinician spends on the participant giving guidance through telephone calls and/or written guidance, in minutes, lower is better

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Psychiatry Research, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD available anonymized on reasonable request.

REFERENCES:
- [Derived] Hentati A, Hentati Isacsson N, Rosen A, Jernelov S, Kaldo V, Ljotsson B, Forsell E, Lindefors N, Kraepelien M. Effects of intervention design on engagement and outcomes in digital self-help for insomnia - factorial RCT. NPJ Digit Med. 2025 Jul 8;8(1):416. doi: 10.1038/s41746-025-01839-0. PMID 40628992